CLINICAL TRIAL: NCT03394040
Title: Point-of-Use Pathogen Identification Tool for Diarrhea
Status: Terminated | Type: Observational
Why Stopped: PI left the NIH
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180040; 18-NR-0040
Record Dates: First submitted 2018-01-05; First posted 2018-01-09 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Diarrhea
Keywords: Diarrhea; Point-of-Need; Pathogen Identification
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: The study seeks individuals of all ages experiencing diarrhea from the Washington Metropolitan area

SUMMARY:
Background:

Many people suffer from diarrhea every year. In the United States, it leads to about 130,000 hospitalizations and 3,000 deaths a year. Researchers want to test a tool that may show them what germs cause diarrhea. It is a simple paper strip test and doesn t require electric power. This may make it easier for health care workers to more quickly fight diarrheal diseases.

Objective:

To test a tool that may detect what germs cause diarrhea.

Eligibility:

People already enrolled in an active NIH protocol who have diarrhea

Design:

Participants will have 1 or 2 studies. They will give information about their symptoms, current medicines, and basic personal data. They will give a stool sample.

Part of each sample will be tested in a lab. The rest will be stored indefinitely. No personal data will be connected to the samples. The stored samples may be used in future research.

Positive test results will be reported to a participant s primary doctor

DETAILED DESCRIPTION:
Objective

This is a cross-sectional study to validate a new, simple, rapid and affordable point-of-use pathogen identification research tool (hence forth referred to as the "tool") of diarrheal diseases for potential use in resource limited settings in the future. The tool was developed under the terms of a National Institutes of Health (NIH) approved Clinical CRADA between NINR and GoDx, Inc. The sensitivity and specificity of the tool in identifying several common gastrointestinal (GI) pathogens in stool will be examined in participants with diarrhea. The proposed validation study will constitute the initial assessment of the tool in a healthcare environment. Once the detection validity and technical performance of the tool have been evaluated in this context, the tool will be further tested in low resource healthcare settings.

Study population

Study participants will be recruited from the Washington, DC, metropolitan area using standard NIH recruitment practices, as well as from among participants in two existing protocols (09-NR-0064, 12-NR-0195) which recruit and consent research participants with GI disorders and diseases. Lastly, participants enrolled on other NIH protocols will be recruited. Appropriate stool samples may also be sequestered from an exempt repository protocol (09-NR-N228). All ages, ethnicities and both sexes will be considered for inclusion in this study. The study population would reflect the demographics of the greater Washington DC metropolitan area. Externally recruited participants and participants recruited from existing protocols will be asked to supply stool samples. A total of 800 samples from participants with diarrhea will be included in this study.

Design

Stool samples will be collected from participants with diarrhea for which pathogen testing using the NIH standard of care, BioFire FilmArray GI Pathogen Panel (FDA approved PCR based pathogen diagnostic) by the Department of Laboratory Medicine (DLM) is indicated. Collected stool samples will be tested for pathogens causing GI disease, using the FilmArray GI panel by the DLM. Technicians in the NINR laboratories will test aliquots from the same stool samples using our tool. The tool has been designed for detection of the most common diarrhea causing pathogens. Of primary interest for this study are: Enteropathogenic Escherichia coli - EPEC, Clostridium difficile C. difficile, Enteroaggregative Escherichia coli - EAEC, and Campylobacter spp. Pathogens of secondary interests, but for which the study is not specifically powered, will also be included and are: Shigella sp., Shiga Toxin-Producing Escherichia coli - STEC, Salmonella spp., and Cryptosporidium spp. Participants will not receive results from the tool.

Outcome measures

The percent sensitivity (ability to make the correct positive identification), specificity (ability to make the correct negative identification) and 95% confidence intervals will be statistically determined by comparing the results yielded by the tool and the FilmArray GI panel. Controlled laboratory experiments suggest >90% specificity and sensitivity of the tool for the detection of the specified pathogens.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. We will include samples from participants with self-reported or clinical provider documented diarrhea defined as one or more loose or watery stools per day as defined by criteria a or b below:

     * Cases of acute diarrhea (i.e., diarrhea which is currently active or was experienced up to one day prior to sampling or still active during sampling) will be included.
     * Cases of persistent diarrhea (i.e., diarrhea which is chronic or chronic-intermittently, i.e., once a week or more, experienced for at least 2 to 4 weeks prior to sampling), will be included. In the case of chronic diarrhea, diarrhea does not have to be active on the day of, or immediately prior to (i.e., one day) sampling.
  2. Current enrollment in an active NIH protocol or enrollment in 12-NR-0195.
  3. Able to provide 50ml stool sample within 2-3 hours.
  4. Children will only be enrolled if they are currently enrolled in an active NIH protocol or enrolled in 12-NR-0195.

EXCLUSION CRITERIA:

1. This protocol will exclude outpatients who are clinically unstable patients. Clinically unstable patient is defined as someone requiring emergent care or hospitalization.
2. Antibiotic use, which can affect intestinal flora, is not exclusionary but will be controlled for via post-hoc analysis.
3. NINR employees, subordinates/relatives/ or co-workers.
4. Any NIH employee who is a subordinates/relatives/or co-workers of study investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study seeks individuals of all ages experiencing diarrhea from the Washington Metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to validate the tool in detecting diarrhea causing pathogens in stool. The sensitivity and specificity of the tool to identify the common diarrhea causing pathogens in the US. | At enrollment
  The study aims to validate the tool in detecting pathogens that cause diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A Henderson, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-NR-0040.html